CLINICAL TRIAL: NCT00073762
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Two Fixed Doses (200 Mg, Or 400 Mg) Of DVS-233 SR In Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 SR In Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-308?
Record Dates: First submitted 2003-12-04; First posted 2003-12-08 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
Primary Objective: To compare the antidepressant efficacy and safety of subjects receiving DVS-233 SR versus subjects receiving placebo.

Secondary Objective: To assess the response of subjects receiving DVS-233 SR for the clinical global evaluation, functionality, general wellbeing, pain, and absence of symptoms (Hamilton Psychiatric Rating Scale for Depression, 17-item [HAM-D17] less than or equal to 7) versus those subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Sexually active women participating in the study must use a medically acceptable form of contraception
* Subjects must have a primary diagnosis of major depressive disorder of 4 on Clinical Global Impressions-Severity scale (CGI-S)

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past
* Treatment with venlafaxine (immediate release [IR] or extended release [ER]) within 90 days of study day 1
* Known hypersensitivity to venlafaxine (IR or ER)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058